CLINICAL TRIAL: NCT06478589
Title: Patient Priorities for Survivorship Care in Older Breast Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dana Giza, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-23-0591; K12TR004908-02 (NIH); 1R03AG089057-01 (NIH)
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Survivorship
Keywords: Patient priorities; Survivorship Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Patient Priorities Care (PPC) approach plus Usual Care (Experimental): Older adults breast cancer survivors will have a visit with a facilitator to discuss about their health priorities for breast cancer survivorship care prior to their usual visit with the oncology/primary care physicians to discuss about aspects of survivorship care
  Interventions: Behavioral: Adapted Patient Priorities Care (PPC) approach; Other: Usual Care
- Usual Care (Active Comparator): Older adults breast cancer survivors will have usual healthcare visits with the oncology/primary care physicians to discuss aspects of survivorship care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Adapted Patient Priorities Care (PPC) approach — Step 1 is a PPC facilitation encounter, at which the facilitator will help the participant identify patient priorities, such as clarifying values (what matters most); setting meaningful, specific, and realistic outcome goals; describing healthcare preferences (care that is helpful and/or burdensome) and tradeoffs; and discussing priorities with clinicians. The participant's healthcare priorities are then documented and transmitted to clinicians, in order to facilitate changes in the patient's care plan to align it with his/her priorities. In step 2, the clinician considers patient's priorities and potential healthcare options (options might include starting or stopping treatments; adding or removing medications; ordering more or fewer tests; recommending or removing self-management tasks). In step 3, the clinician discusses care options with the participant, using strategies for aligning care with patient priorities.
  Arms: Adapted Patient Priorities Care (PPC) approach plus Usual Care
Other: Usual Care — Usual care for breast cancer survivorship includes regular visits with the oncology provider and yearly mammograms for surveillance.

SUMMARY:
The objective of this study is to adapt the Patient Priorities Care (PPC) framework to breast cancer survivorship via a user-centered approach, through an iterative process in which patients and their physicians help to refine and modify the intervention. A second objective is to evaluate the feasibility and effectiveness of the adapted PPC framework in breast cancer survivorship for older adults.

DETAILED DESCRIPTION:
In the proposed project, we will use a Patient Priorities Care framework to explore older breast cancer survivors' priorities and health care preferences for high-quality breast cancer survivorship. The framework will include two components: (1) a health priorities identification session with a facilitator, and (2) an encounter with the oncology provider to discuss changes in the patient's care plan to align it with his/her priorities. Our overall hypothesis is that prioritizing patients' priorities is feasible and facilitates individualized survivorship care for older women with breast cancer and multiple chronic conditions. An advisory panel composed of oncologists, geriatricians, and patient advocates will provide regular feedback throughout the refinement and adaptation of the Patient Priorities Care framework to the breast cancer survivorship context and engage in an iterative process of development. After incorporating feedback from the stakeholder panel to create an adapted version of the framework, we will carry out a randomized quality improvement project with the objective of evaluating the feasibility of using the framework in the context of breast cancer survivorship and provide empirical estimates of treatment effect sizes by measuring treatment burden and quality of life at 3 months, adherence to basic and priorities driven survivorship care recommendations at 12 months. Ultimately, the results of this project will provide initial direction for intended improvement, which will be verified in a larger, future trial.

ELIGIBILITY:
Inclusion Criteria:

* able to write and speak English
* Stage DCIS/I/II/III breast cancer diagnosis
* 3 months from active cancer therapy (including first or second-line treatment chemotherapy, radiation and/or surgery, or multimodal treatment) up to 10 years since completing treatment
* ≥3 documented comorbidities by chart review, or taking ≥10 medications, have ≥ 1 hospitalization over the past year, ≥ 2 emergency department visits over the past year, seen by > 2 specialists over the past year
* able to provide consent

Exclusion Criteria:

* currently on active cancer therapy (including first or second-line treatment chemotherapy, radiation and/or surgery, or multimodal treatment)

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment burden as assessed by the treatment burden questionnaire (TBQ) | baseline
  The treatment burden questionnaire (TBQ) measures perceptions of burden of overall care (for example, medication taking, self monitoring, visits to the provider, tests, tasks to access and coordinate care). Total score ranges from 0 to 150, and a higher score indicates greater perceived burden.
Treatment burden as assessed by the treatment burden questionnaire (TBQ) | 3 months
  The treatment burden questionnaire (TBQ) measures perceptions of burden of overall care (for example, medication taking, self monitoring, visits to the provider, tests, tasks to access and coordinate care). Total score ranges from 0 to 150, and a higher score indicates greater perceived burden.
Treatment burden as assessed by the treatment burden questionnaire (TBQ) | 6 months
  The treatment burden questionnaire (TBQ) measures perceptions of burden of overall care (for example, medication taking, self monitoring, visits to the provider, tests, tasks to access and coordinate care). Total score ranges from 0 to 150, and a higher score indicates greater perceived burden.
Health status as assessed by the Functional Assessment of Cancer Therapy - Breast (FACT-B) | baseline
  The Functional Assessment of Cancer Therapy- Breast (FACT-B) is a standardized approach to objectively evaluate and quantify the overall health status of patients with subscales measuring physical, social, emotional, and functional well-being. Total score ranges from 0 to 148, where a higher score indicates a better outcome.
Health status as assessed by the Functional Assessment of Cancer Therapy - Breast (FACT-B) | 3 months
  The Functional Assessment of Cancer Therapy- Breast (FACT-B) is a standardized approach to objectively evaluate and quantify the overall health status of patients with subscales measuring physical, social, emotional, and functional well-being. Total score ranges from 0 to 148, where a higher score indicates a better outcome.
Health status as assessed by the Functional Assessment of Cancer Therapy - Breast (FACT-B) | 6 months
  The Functional Assessment of Cancer Therapy- Breast (FACT-B) is a standardized approach to objectively evaluate and quantify the overall health status of patients with subscales measuring physical, social, emotional, and functional well-being. Total score ranges from 0 to 148, where a higher score indicates a better outcome.

SECONDARY OUTCOMES:
Number of participants who adhere to survivorship basic recommendations | from baseline to 12 months
  Survivorship basic recommendations for breast cancer survivors, as recommended by the American Society of Clinical Oncology (ASCO) guidelines, include receiving a detailed cancer-related history and physical examination every 3-6 months for the first 3 years and every 6 to 12 months for the next 2 years, as well as having an annual mammogram (unilateral if for unilateral mastectomies or bilateral for patients with lumpectomies or other breast conserving strategies).
Number of participants who adhere to priorities-driven survivorship recommendations | from baseline to 12 months
  Adherence to priorities-driven survivorship recommendations will focus on adherence to medications, self-management tasks, procedures, tests or referrals recommended during survivorship care based on patient's priorities.

CONTACTS AND LOCATIONS:
Overall Officials: Dana E. Giza, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - UT Physicians Center for Healthy Aging Bellaire, Bellaire, Texas
  - UT Physicians Family Medicine Bayshore, Houston, Texas
  - Memorial Hermann Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No